CLINICAL TRIAL: NCT01550120
Title: Free Fatty Acids: Threshold Repeatability Study
Status: Completed | Type: Observational
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Richard Mattes, Distinguished Professor, Purdue University
Other Study IDs: 055-027
Record Dates: First submitted 2012-03-07; First posted 2012-03-09 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-03

CONDITIONS: Taste, Non-esterified Fatty Acids
Keywords: taste; fat; threshold; sensitivity; human
MeSH Terms: conditions — Platelet Glycoprotein IV Deficiency; Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study seeks to determine if non-esterified fatty acid (NEFA) taste detection thresholds change with repeated testing. Threshold testing for NEFA taste has been reported by a number of laboratories, including our own; however, these studies have reported data for only one testing occasion. The investigators seek to conduct repeated testing to measure the test-retest reliability of these methods. The investigators believe that with repeated exposure to NEFA, a person's sensitivity increases. The investigators are also testing the efficiency of testing by two methods (forced-choice ascending trial versus staircase). Additionally, the association between taste responses, diet and BMI will be explored.

ELIGIBILITY:
Inclusion Criteria:

* 18-55 years old
* in good health
* available for three months

Exclusion Criteria:

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants between the ages of 18 and 55 years of age from any ethnic background who are in good health and are available for the next three months will be recruited. Additionally, equal numbers of lean and overweight participants will be sought.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2012-03; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Non-esterified fatty acid detection thresholds in humans | 6 months
BMI | Baseline

SECONDARY OUTCOMES:
Habitual fat intake | Baseline
  Block Rapid Dietary Fat Screener will be used as well as the ASA-24.
testing method | 6 months
  Comparison of time to maximum sensitivity by participants based on forced-choice versus staircase stimulus presentation techniques.
hunger | each visit
  Visual analog scale

CONTACTS AND LOCATIONS:
Overall Officials: Richard D Mattes, PhD, Principal Investigator — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States